CLINICAL TRIAL: NCT04696237
Title: National Treatment Approach Versus Standardized Treatment Protocol to Manage Patients With Cleft Lip and Palate: a Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hana Adel Adawy, Resident in the Department of Orthodontics, Cairo University
Other Study IDs: HanaAdelAdawyCU2021
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (9):
- orthodontists: orthodontists with more than 2 years of working experience
  Interventions: Other: Questionnaire
- general dentists: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- oral and maxillofacial surgeons: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- plastic surgeons: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- cleft nurses: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- speech therapists: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- ENT specialists: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- psychiatrists: with more than 2 years of working experience
  Interventions: Other: Questionnaire
- Social workers: with more than 2 years of working experience

INTERVENTIONS:
Other: Questionnaire — a questionnaire to provide data about the management of cleft lip and palate patients in Egypt will be designed
  Groups: ENT specialists; cleft nurses; general dentists; oral and maxillofacial surgeons; orthodontists; plastic surgeons; psychiatrists; speech therapists

SUMMARY:
The main objective of this study is to provide data about treatment protocols for CLP patients in Egypt, and compare it to the management protocol suggested by the ACPA.

DETAILED DESCRIPTION:
This is a cross-setional survey to gather data concerning the current CL/P situation in our country.

The main objectives of this study are

1. To identify if the healthcare providers in Egypt work in cleft centers or teams
2. To assess if the healthcare providers are aware of the interdisciplinary team-based treatment approach that should be followed for CLP patients' management.
3. To provide data about the cleft lip and palate management protocols that are being followed in Egypt.
4. Evaluation of the current status of cleft care and experiences of the health care providers involved in the management of the CLP in Egypt including Orthodontists, OMFS, Otolaryngologists, Plastic Surgeons, Speech therapists, Dentists, Psychiatrists, Psychologists, Pediatricians, Nurses and Social Workers.
5. Identify the presence or absence of cleft centers in our country.
6. Identify the presence or absence or organized healthcare services for the CLP patients in terms of parents' awareness about the condition and its management, as well as the presence of medical referrals between the specialists.
7. Reporting the patients/parents' experiences throughout their treatment journey.
8. Highlight the obstacles that could be faced by the health care providers as well as the patients along the treatment journey.

ELIGIBILITY:
Inclusion Criteria:

* • A sample of CLP patients of varying age groups: (Neonate and Infant (Birth -2 years of age), Primary Dentition Stage (2 to 6 Years of Age), Permanent Dentition Stage)

  * CLP patients' parents will be included to answer questions involving CLP infants and adolescents
  * Paediatric dentists
  * Paediatricians
  * GP dentists
  * Oral and maxillofacial surgeons
  * Plastic surgeons
  * Orthodontists
  * Nurses
  * Speech therapists
  * Prosthodontists
  * Psychiatrists
  * Psychologists
  * Social workers
  * Otolaryngologists

Exclusion Criteria:

* patients who don't suffer from cleft lip and palate
* other specialists who aren't involved in the CLP team

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all the specialists involved in the management of cleft lip and palate patients as well as cleft lip and palate adult patients will be involved in the questionnaire
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
the presence or absence of a multidisciplinary treatment approach for CLP patients | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CairoU, Cairo, Egypt